CLINICAL TRIAL: NCT01968681
Title: Treatment of Nevus Flammeus With Alexandrite Laser
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bispebjerg Hospital (Other)
Responsible Party: Principal Investigator, Merete Haedersdal, Professor, Bispebjerg Hospital
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: H-4-2013-066
Record Dates: First submitted 2013-10-21; First posted 2013-10-24 (Estimated); Last update posted 2015-02-24 (Estimated); Status verified 2015-02

CONDITIONS: Nevus Flammeus
MeSH Terms: conditions — Port-Wine Stain | interventions — Lasers, Solid-State

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- Alexandrite laser treatment (Experimental)
  Interventions: Procedure: Alexandrite laser

INTERVENTIONS:
Procedure: Alexandrite laser — 3 different alexandrite laser settings are used in respectively 3 different treatment areas and compared with a non-treated control area.
  Other Names: Candela Gentle Max

SUMMARY:
Nevus flammeus is a congenital vascular malformation. Nevus flammeus is traditionally treated with pulsed dye lasers (PDL); however, around 20 percent of patients are poor responders and do not get satisfactory results from pulsed dye laser treatments.

Small studies with alexandrite lasers indicate that this may be an alternative treatment for individuals with nevus flammeus. This study assesses the clinical effect and side effects of alexandrite laser treatment for nevus flammeus using different treatment settings.

ELIGIBILITY:
Inclusion Criteria:

* 10 or more years of age
* Fitzpatrick Skin Type I-III
* Previously untreated or pulsed dye laser-insufficiently treated nevus flammeus
* Nevus flammeus size minimum 8 x 2 centimeter within one anatomical region
* Written and oral informed consent

Exclusion Criteria:

* Known light sensibility toward visible light
* Tendency to develop hypertrophic scars or keloids
* Fitzpatrick Skin Type IV-VI
* Individuals, that are obviously pigmented due to recent sun exposure or sun beds
* Treatment with systemic retinoids within 6 months
* Pregnancy and lactation
* Unwillingness to complete protocol

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2013-09; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Reduction in clinical appearance on a 10-point scale | 6-8 weeks

SECONDARY OUTCOMES:
Skin reflectance measurement to assess degree of redness | 6-8 weeks
Skin reflectance to assess degree of pigmentation | 6-8 weeks

OTHER OUTCOMES:
Clinical assessment of pigmentation | 6-8 weeks
Clinical assessment of scar tissue formation | 6-8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Merete Haedersdal, Professor, Principal Investigator — Bispebjerg Hospital
Locations (1):
- Bispebjerg Hospital, Copenhagen, Denmark